CLINICAL TRIAL: NCT03297060
Title: Implementing Alcohol Misuse SBIRT in a National Cohort of Pediatric Trauma Centers
Acronym: IAMSBIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R01AA025914 (NIH); 1R01AA025914 (NIH)
Record Dates: First submitted 2017-09-08; First posted 2017-09-29 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2023-11

CONDITIONS: Alcohol Drinking
Keywords: Alcohol Screening
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This study utilizes a stepped wedge design.
Who Masked: Participant
Masking Description: Participants will not know which arm their institution has been assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SSL Implementation Strategy (Experimental): Science to Service Implementation Strategy for SBIRT adherence
  Interventions: Other: SSL Implementation Strategy
- Standard Care (No Intervention): Standard Care SBIRT services

INTERVENTIONS:
Other: SSL Implementation Strategy — Science to Service Laboratory (SSL) is an approach developed by the SAMHSA-funded Addiction Technology Transfer Centers (ATTCs) that consists of didactic training + performance feedback + leadership coaching to improve SBIRT adherence within the pediatric trauma center
  Arms: SSL Implementation Strategy

SUMMARY:
The goal of this study is to conduct a fully powered Type III hybrid effectiveness-implementation trial to test the effectiveness of a comprehensive implementation strategy in increasing the implementation of SBIRT for alcohol and other drug use in pediatric trauma centers. Our implementation strategy is based on the Science to Service Laboratory (SSL), an approach developed by the SAMHSA-funded Addiction Technology Transfer Centers (ATTCs) that consists of the same three core elements (i.e., didactic training + performance feedback + leadership coaching) used in our Centers for Disease Control and Prevention (CDC) study. Based on feedback from the CDC study, two enhancements were made to the SSL strategy: 1) integration of the intervention into the electronic medical record as a means of improving SBIRT adherence; and 2) development of separate training tracks for nurses, social workers and organizational leaders to meet the unique needs of each group. In addition, we integrate counseling around the use of prescription pain relievers into the SBIRT intervention as an Exploratory Aim, since most pediatric trauma center patients are discharged on pain medication and patients with a history of AOD use are at elevated risk of opioid misuse. Utilizing a stepped wedge design, a national cohort of 10 pediatric trauma centers will receive the SSL implementation strategy. Data collection for this study relies on multiple sources. At six distinct time points, each of the 10 sites will provide retrospective data from EMR charts. A subset of adolescents will also report on fidelity of intervention delivery and linkage to care (i.e., continued AOD discussion and/or treatment with a primary care provider) 1 month post hospital discharge. In addition, nurses, social workers, and leaders from each pediatric trauma center will report on organizational readiness for implementation at three distinct time points. Results of this study will demonstrate that a highly scalable implementation strategy, adapted for pediatric trauma centers from the results of our mixed-methods implementation trial, will improve the fidelity (i.e., the consistency and quality) of SBIRT delivery in pediatric trauma centers.

DETAILED DESCRIPTION:
In 2006, the American College of Surgeons (ACS) adopted a requirement for certification as a level one trauma center that mandated universal screening for alcohol misuse and delivery of a brief intervention for those screening positive1. Though this requirement has been mandated for a decade, its implementation has been challenging, especially for pediatric trauma centers. Our research team completed a CDC funded implementation study supporting seven pediatric trauma centers' compliance with the ACS requirement by developing and implementing an institutional alcohol Screening, Brief Intervention and Referral to Treatment (SBIRT) protocol for adolescent trauma patients. A mixed-methods approach indicated that SBIRT adoption rates increased at all sites2; however, providers' fidelity to the SBIRT intervention was variable, and providers reported a number of barriers to SBIRT implementation. We have an unparalleled opportunity and an identified need to evaluate the effectiveness of a comprehensive SBIRT implementation strategy for alcohol and other drug (AOD) use across a national cohort of pediatric trauma centers.

The goal of this application is to conduct a fully powered Type III hybrid effectiveness-implementation trial to test the effectiveness of a comprehensive strategy in improving the implementation of SBIRT for AOD use in pediatric trauma centers. Our implementation strategy is based on the Science to Service Laboratory (SSL), an approach developed by the SAMHSA-funded Addiction Technology Transfer Centers (ATTCs) that consists of the same three core elements (i.e., didactic training + performance feedback + leadership coaching) used in our CDC study. The SSL is an evidence-based strategy3,4 that provides leadership coaching focused on sustainability and that has potential for widespread dissemination throughout the ATTC network. The SSL was specifically designed to increase organizational readiness for implementation. Based on feedback from the CDC study, two enhancements were made to the SSL strategy: 1) integration of the intervention into the electronic medical record (EMR) as a means of improving SBIRT adherence; and 2) development of separate training tracks for nurses, social workers and organizational leaders to meet the unique needs of each group. In addition, we integrate counseling around the use of prescription pain relievers into the SBIRT intervention as an Exploratory Aim, since most pediatric trauma center patients are discharged on pain medication and patients with a history of AOD use are at elevated risk of opioid misuse5. Utilizing a stepped wedge design, a national cohort of 10 pediatric trauma centers will receive the SSL implementation strategy. Data collection for this study relies on multiple sources. At six distinct time points, each of the 10 sites will provide retrospective data from EMR charts for review. A subset of adolescents will also report on fidelity of intervention delivery and linkage to care (i.e., continued AOD discussion and/or treatment with a primary care provider) 1 month after hospital discharge. In addition, nurses, social workers, and leaders from each pediatric trauma center will report on organizational readiness for implementation at three distinct time points. Results of this study will demonstrate that a highly scalable implementation strategy, adapted for pediatric trauma centers from the results of our mixed-methods implementation trial, will improve the fidelity (i.e., the consistency and quality) of SBIRT delivery within pediatric trauma centers.

Primary Aim: Evaluate the effectiveness of the SSL implementation strategy in increasing fidelity of SBIRT delivery at pediatric trauma centers, relative to usual implementation.

Hypothesis: Staff that receive the SSL will increase by 20% the proportion of admitted injured adolescents receiving each element of the SBIRT protocol as indicated: a) validated AOD screening, b) brief AOD intervention, and c) referral to appropriate care post-discharge (i.e., continued AOD discussion/treatment with a health care provider).

Secondary Aim 1: Evaluate whether readiness for organizational change mediates the influence of the SSL implementation strategy on implementation effectiveness (i.e., fidelity of SBIRT delivery).

Hypothesis: The effect of the SSL on implementation effectiveness will be partially mediated by organizational readiness to change.

Secondary Aim 2: Evaluate the effect of the SSL implementation strategy on improving patient linkage to appropriate care (i.e., continued AOD discussion with primary care provider and/or AOD treatment) following discharge from pediatric trauma centers.

Hypothesis: Injured adolescents that receive the SSL will report higher rates of AOD discussion/treatment with a health care provider within 30 days of discharge, compared to usual implementation.

Exploratory Aim: Examine the integration of counseling regarding the use of prescription pain relievers into SBIRT delivery with injured adolescent patients who screen positive for AOD use.

Hypothesis: Staff that receives the SSL will demonstrate higher rates of discussion of appropriate pain medication use and medication disposal with patients who screen positive for AOD use, compared to usual implementation.

The proposed research builds on our prior implementation research and has potential to impact clinical care, address an important public health issue and significantly contribute to implementation science.

ELIGIBILITY:
Inclusion Criteria: Eligible adolescents must meet these criteria:

12-17 years of age Admitted to a participating trauma service for an injury Screened positive for AOD use based on biologic testing or self-report on the alcohol screening tool (S2BI) Fluent in English Able to provide written assent and parent able to provide written consent.

Exclusion Criteria: Exclusion criteria include:

Prisoner or in police custody Admitted due to suicide attempt Any acute conditions that would preclude provision of informed consent (i.e., acute psychosis, altered mental status, cognitive impairment).

-

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 430 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Proportion of admitted injured adolescents receiving each element of the alcohol screening, brief intervention and referral to treatment (SBIRT) protocol | 54 months
  SBIRT components will be collected through retrospective data abstraction of each site's electronic medical record to determine if admitted injured adolescent patients received the SBIRT components during the different phases of the study.

SECONDARY OUTCOMES:
Rate of readiness for organizational change within each institution | 9 months
  Participating staff will complete organizational readiness for implementing change surveys throughout the study to identify if organizational readiness to change mediates implementation effectiveness
Percent of adolescents with screened positive for AOD use and who reported linkage to discussions about AOD with a health care provider within 30 days of discharge within 30 days of discharge | 30 days
  Patients will complete an online survey 30 days after discharge to determine linkage to appropriate care( i.e., continued AOD discussion with primary care provider and/or AOD treatment) following discharge from pediatric trauma centers.)

OTHER OUTCOMES:
Rate of discussion of appropriate pain medication use and medication disposal with patients who screen positive for alcohol or other drug use. | 9 months
  Rates will be determined through EMR review (rates of documented opioid counseling).

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Mello, MD, MPH, Principal Investigator — Rhode Island Hospital
Locations (1):
- Rhode Island Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Scott K, Mello MJ, Almonte G, Lemus EA, Bromberg JR, Baird J, Spirito A, Zonfrillo MR, Lawson K, Lee LK, Christison-Lagay E, Ruest S, Aidlen J, Kiragu A, Pruitt C, Nasr I, Maxson RT, Ebel B, Becker SJ. A qualitative process evaluation of SBIRT implementation in pediatric trauma centers using the Science to Service Laboratory implementation strategy. Implement Sci Commun. 2025 Jan 30;6(1):13. doi: 10.1186/s43058-025-00697-x. PMID 39885597
- [Derived] Mello MJ, Baird J, Spirito A, Scott K, Zonfrillo MR, Lee LK, Kiragu A, Christison-Lagay E, Bromberg J, Ruest S, Pruitt C, Lawson KA, Nasr IW, Aidlen JT, Maxson RT, Becker S. Adolescents' Perceptions of Screening, Brief Intervention, and Referral to Treatment Service at Pediatric Trauma Centers. Subst Use. 2024 Aug 21;18:29768357241272356. doi: 10.1177/29768357241272356. eCollection 2024 Jan-Dec. PMID 39175910
- [Derived] Mello MJ, Lee LK, Christison-Lagay E, Spirito A, Becker S, Bromberg J, Ruest S, Zonfrillo MR, Scott K, Pruitt C, Lawson K, Nasr I, Aidlen J, Baird J. Counseling for opioids prescribed at discharge of hospitalized adolescent trauma patients. Inj Epidemiol. 2023 Oct 23;10(Suppl 1):53. doi: 10.1186/s40621-023-00465-2. PMID 37872639
- [Derived] Mello MJ, Baird J, Bromberg JR, Spirito A, Zonfrillo MR, Lee LK, Christison-Lagay ER, Ruest SM, Pruitt CW, Lawson KA, Kiragu AW, Nasr I, Aidlen JT, Ebel BE, Maxson RT, Scott K, Becker SJ. Variability in opioid pain medication prescribing for adolescent trauma patients in a sample of US pediatric trauma centers. Trauma Surg Acute Care Open. 2022 Apr 26;7(1):e000894. doi: 10.1136/tsaco-2022-000894. eCollection 2022. PMID 35558645
- [Derived] Mello MJ, Becker SJ, Spirito A, Bromberg JR, Wills H, Barczyk A, Lee L, Pruitt C, Ebel BE, Zonfrillo MR, Nimaja E, Scott K, Kiragu A, Nasr IW, Aidlen JT, Maxson RT, Baird J. Screening Adolescent Trauma Patients for Substance Use at 10 Pediatric Trauma Centers. J Trauma Nurs. 2020 Nov/Dec;27(6):313-318. doi: 10.1097/JTN.0000000000000537. PMID 33156244
- [Derived] Mello MJ, Becker SJ, Bromberg J, Baird J, Zonfrillo MR, Spirito A. Implementing Alcohol Misuse SBIRT in a National Cohort of Pediatric Trauma Centers-a type III hybrid effectiveness-implementation trial. Implement Sci. 2018 Feb 22;13(1):35. doi: 10.1186/s13012-018-0725-x. PMID 29471849

DOCUMENTS (1):
  • Informed Consent Form (2021-04-26): https://cdn.clinicaltrials.gov/large-docs/60/NCT03297060/ICF_003.pdf